CLINICAL TRIAL: NCT06509113
Title: Reducing Stigmatizing Attitudes and Behaviors of Nursing Students in Simulated Clinical Visits of Patients Living With HIV in Iran
Brief Title: A Pilot Study of an Online HIV Stigma Training for Nursing Students in Iran
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ponce Health Sciences University (Other); Kerman University of Medical Science (Unknown); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-38482; R01TW012408 (NIH)
Record Dates: First submitted 2024-07-02; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Stigma, Social; HIV Infections
Keywords: Stigma; HIV; Training; Iran; Student; Nursing
MeSH Terms: conditions — Social Stigma; HIV Infections

STUDY DESIGN:
Intervention Model Description: The investigators will develop a 4-module online HIV stigma reduction training with simulated patients for nursing students in the intervention arm. This training includes three case scenarios: a male who injects drugs, a male who has sex with men, and a female sex worker, all with HIV. Interviews with people living with HIV (PLWH) and focus groups with nursing students and faculty will refine the content. The control group will receive a course on HIV epidemiology without stigma-specific content. To assess efficacy, 70 nursing students will initially have a clinical encounter with a simulated patient on a non-HIV topic. A week later, they will have an HIV visit and complete stigma and empathy scales. Participants will then be randomized into two groups: one receiving stigma training and the other, HIV epidemiology training. Afterward, they will have another HIV-related clinical encounter and complete the scales again.
Masking Description: To avoid potential bias based on the timing of enrollment, The investigators will use "block randomization" with randomly permuted block sizes to avoid identification of the allocation of the last participant in a block. Once a nursing student completes their baseline stigma and empathy survey, participants will be assigned the next masked envelope from the randomization list by a research staff, which in turn assign the person to one of the two study arms. The research staff and participants are masked to study arm assignment prior to opening the envelopes. The person analyzing the data will be masked to study arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Nursing students will be assigned to the intervention group and will receive online HIV-related stigma training.
  Interventions: Behavioral: The online HIV-related stigma training
- Control (Other): Nursing students will be assigned to the online HIV epidemiology training with no specific content on stigma.
  Interventions: Behavioral: The online HIV epidemiology training with no specific content on stigma

INTERVENTIONS:
Behavioral: The online HIV-related stigma training — The intervention is an online HIV-related stigma training that takes 6 hours in 4 weeks to be completed.
  Arms: Intervention
Behavioral: The online HIV epidemiology training with no specific content on stigma — Nursing students will be trained in an online HIV epidemiology training with no specific content on stigma. It will take 6 hours in 4 weeks to complete the training.
  Arms: Control

SUMMARY:
In this study, the investigators will assess the feasibility, acceptability, and preliminary efficacy of online HIV stigma training in reducing stigmatizing attitudes and behaviors of nursing students in simulated clinical visits of patients living with HIV compared to an online HIV epidemiology training with no specific content on stigma.

DETAILED DESCRIPTION:
Iran has the highest burden of HIV in the Middle East. However, only 42% of Iranians living with HIV are diagnosed and 28% on antiretroviral therapy. The largest gap in the continuum of HIV care is diagnosis. Due to sociocultural and religious beliefs, HIV- associated stigma and drug use stigma are exceedingly high, and sex outside of marriage, or sex of man with another man are considered to be "sinful" behaviors. These intersectional stigmas (stigma towards drug use, sexism, and homophobia) in addition to HIV stigma are major barriers for many people at risk for or living with HIV to engage in HIV testing or treatment. Our prior studies found that health providers have limited clinical encounters with people living with HIV (PLWH) and have no HIV stigma training. This lack of training can lead to stigmatizing attitudes and behaviors towards people at risk for HIV or PLWH. The highest HIV stigmatizing behaviors was reported in nurses and physician assistants. These data, coupled with the extreme marginalization of key populations at high risk for HIV in Iran, call for the development of new ways to train nurses to reduce HIV-related stigma in clinical settings. The investigators propose to develop, and field test an HIV stigma online training including simulated patients living with HIV for nursing school students. In a randomized controlled trial, the investigators will assess the feasibility, acceptability, and preliminary efficacy of the online HIV stigma training in reducing stigmatizing attitudes and behaviors of nursing students in simulated clinical visits of patients living with HIV compared to an online HIV epidemiology training with no specific content on stigma. Successful development of the HIV stigma training and simulated patients at risk for or living with HIV will set the stage for developing a larger trial of nurses and other health providers which can lead to an effective and scalable training program to reduce HIV-related stigma in clinical settings and improve engagement in HIV testing and care services. The investigators from the University of California San Francisco (UCSF), will lead and co-investigate the project, respectively. They will collaborate with teams from Kerman University of Medical Sciences (KMU), Iran, and Ponce Health Sciences University (PHSU) in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Currently nursing students in their year 3 or 4 of training
* Kerman Medical University (KMU) nursing schools

Exclusion Criteria:

* Nursing student in their year 1 and 2
* Students of other fields and other universities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stigma score | Up to 4 weeks before and after intervention
  All nursing students will complete a validated stigma scale before and after the training interventions.
Behavioral manifestations of HIV stigma | Up to 4 weeks before and after intervention
  Before and after the training interventions, all nursing students will meet with a randomly selected simulated patient for an HIV visit. These visits will be video recorded and will be coded and scored for stigmatizing behaviors.
Empathy score | Up to 4 weeks before and after intervention
  All nursing students will complete a validated empathy scale before and after the training interventions.

SECONDARY OUTCOMES:
The attitudes and behaviors of nursing students after the online HIV stigma training | Three months after the intervention
  We will qualitatively examine study participants' real-world behaviors with HIV and at-risk patients to (1) explore if behaviors learned during the intervention carry on in real-world settings, (2) better understand how behaviors are manifested in natural settings, and (3) explore best methods to assess behaviors in real-world scenarios

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mirzazadeh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Skill labs at the nursing school of Kerman Medical University, Kerman, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gokengin D, Doroudi F, Tohme J, Collins B, Madani N. HIV/AIDS: trends in the Middle East and North Africa region. Int J Infect Dis. 2016 Mar;44:66-73. doi: 10.1016/j.ijid.2015.11.008. PMID 26948920
- [Background] UNAIDS. Country factsheets Iran 2020. Retrived from https://www.unaids.org/en/regionscountries/countries/islamicrepublicofiran. 2020.
- [Background] Farhoudi B, Ghalekhani N, Afsar Kazerooni P, Namdari Tabar H, Tayeri K, Gouya MM, SeyedAlinaghi S, Haghdoost AA, Mirzazadeh A, Sharifi H. Cascade of care in people living with HIV in Iran in 2019; how far to reach UNAIDS/WHO targets. AIDS Care. 2022 May;34(5):590-596. doi: 10.1080/09540121.2021.1944603. Epub 2021 Jun 28. PMID 34180724
- [Background] Karamouzian M, Akbari M, Haghdoost AA, Setayesh H, Zolala F. "I am dead to them": HIV-related stigma experienced by people living with HIV in Kerman, Iran. J Assoc Nurses AIDS Care. 2015 Jan-Feb;26(1):46-56. doi: 10.1016/j.jana.2014.04.005. Epub 2014 May 2. PMID 24856436
- [Background] Rahmati-Najarkolaei F, Niknami S, Aminshokravi F, Bazargan M, Ahmadi F, Hadjizadeh E, Tavafian SS. Experiences of stigma in healthcare settings among adults living with HIV in the Islamic Republic of Iran. J Int AIDS Soc. 2010 Jul 22;13:27. doi: 10.1186/1758-2652-13-27. PMID 20649967
- [Background] Malekmohammadi N, Mirzazadeh A, Iranpour A, Shafiei Bafti M, Zolala F, McFarland W, et al. HIV Stigma among People Living with HIV in Southeast Iran. Journal of Kerman University of Medical Sciences 2021; 28(5):427-436.
- [Background] Etesam F, Assarian F, Hosseini H, Ghoreishi FS. Stigma and its determinants among male drug dependents receiving methadone maintenance treatment. Arch Iran Med. 2014 Feb;17(2):108-14. PMID 24527971
- [Background] Tavakoli F, Karamouzian M, Rafiei-Rad AA, Iranpour A, Farrokhnia M, Noroozi M, Sharifi A, Marshall BDL, Shokoohi M, Sharifi H. HIV-Related Stigma Among Healthcare Providers in Different Healthcare Settings: A Cross-Sectional Study in Kerman, Iran. Int J Health Policy Manag. 2020 Apr 1;9(4):163-169. doi: 10.15171/ijhpm.2019.92. PMID 32331496
- [Background] Asadi-Aliabadi M, Abolghasemi J, Rimaz S, Majdzadeh R, Rostami-Maskopaee F, Merghati-Khoei E. Barriers to Health Service Utilization Among Iranian Female Sex Workers: A Qualitative Study. J Prev Med Public Health. 2018 Mar;51(2):64-70. doi: 10.3961/jpmph.17.174. PMID 29631351
- [Background] Walker D, Cohen S, Fritz J, Olvera M, Lamadrid-Figueroa H, Cowan JG, Hernandez DG, Dettinger JC, Fahey JO. Team training in obstetric and neonatal emergencies using highly realistic simulation in Mexico: impact on process indicators. BMC Pregnancy Childbirth. 2014 Nov 20;14:367. doi: 10.1186/s12884-014-0367-1. PMID 25409895
- [Background] Walker DM, Cohen SR, Fritz J, Olvera-Garcia M, Zelek ST, Fahey JO, Romero-Martinez M, Montoya-Rodriguez A, Lamadrid-Figueroa H. Impact Evaluation of PRONTO Mexico: A Simulation-Based Program in Obstetric and Neonatal Emergencies and Team Training. Simul Healthc. 2016 Feb;11(1):1-9. doi: 10.1097/SIH.0000000000000106. PMID 26312613
- [Background] Walton A, Kestler E, Dettinger JC, Zelek S, Holme F, Walker D. Impact of a low-technology simulation-based obstetric and newborn care training scheme on non-emergency delivery practices in Guatemala. Int J Gynaecol Obstet. 2016 Mar;132(3):359-64. doi: 10.1016/j.ijgo.2015.08.009. Epub 2015 Dec 11. PMID 26797198
- [Background] Mugo C, Wilson K, Wagner AD, Inwani IW, Means K, Bukusi D, Slyker J, John-Stewart G, Richardson BA, Nduati M, Moraa H, Wamalwa D, Kohler P. Pilot evaluation of a standardized patient actor training intervention to improve HIV care for adolescents and young adults in Kenya. AIDS Care. 2019 Oct;31(10):1250-1254. doi: 10.1080/09540121.2019.1587361. Epub 2019 Feb 27. PMID 30810351
- [Background] Varas-Diaz N, Neilands TB, Cintron-Bou F, Marzan-Rodriguez M, Santos-Figueroa A, Santiago-Negron S, Marques D, Rodriguez-Madera S. Testing the efficacy of an HIV stigma reduction intervention with medical students in Puerto Rico: the SPACES project. J Int AIDS Soc. 2013 Nov 13;16(3 Suppl 2):18670. doi: 10.7448/IAS.16.3.18670. PMID 24242260
- [Background] Varas-Diaz N, Rivera M, Rivera-Segarra E, Neilands TB, Ortiz N, Pedrogo Y, Mendoza S, Rivera Amador A, Martinez Garcia S, Rivera Suazo S, Albizu-Garcia CE. Beyond negative attitudes: Examining HIV/AIDS stigma behaviors in clinical encounters. AIDS Care. 2017 Nov;29(11):1437-1441. doi: 10.1080/09540121.2017.1322679. Epub 2017 May 3. PMID 28464694
- [Background] UNAIDS. Fast-Track: ending the AIDS epidemic by 2030, 2014. Retrieved from https://www.unaids.org/en/resources/documents/2014/JC2686_WAD2014report. 18. UNAIDS. Regional factsheets Middle East and North Africa, 2019. Retrived from https://www.unaids.org/en/regionscountries/middleeastandnorthafrica
- [Background] Feyissa GT, Lockwood C, Woldie M, Munn Z. Reducing HIV-related stigma and discrimination in healthcare settings: A systematic review of quantitative evidence. PLoS One. 2019 Jan 25;14(1):e0211298. doi: 10.1371/journal.pone.0211298. eCollection 2019. PMID 30682131
- [Background] Fahimfar N, Sedaghat A, Hatami H, Kamali K, Gooya M. Counseling and Harm Reduction Centers for Vulnerable Women to HIV/AIDS in Iran. Iran J Public Health. 2013 Jan 1;42(Supple1):98-104. Print 2013. PMID 23865025
- [Background] National AIDS Committee Secretariat, Ministry of Health and Medical Education. Islamic Republic of Iran AIDS progress report on monitoring of the United Nations general assembly special session on HIV and AIDS In; 2017.
- [Background] Sharifi H, Mirzazadeh A, Shokoohi M, Karamouzian M, Khajehkazemi R, Navadeh S, Fahimfar N, Danesh A, Osooli M, McFarland W, Gouya MM, Haghdoost AA. Estimation of HIV incidence and its trend in three key populations in Iran. PLoS One. 2018 Nov 29;13(11):e0207681. doi: 10.1371/journal.pone.0207681. eCollection 2018. PMID 30496204
- [Background] Shahesmaeili A, Karamouzian M, Shokoohi M, Kamali K, Fahimfar N, Nadji SA, Sharifi H, Haghdoost AA, Mirzazadeh A. Symptom-Based Versus Laboratory-Based Diagnosis of Five Sexually Transmitted Infections in Female Sex Workers in Iran. AIDS Behav. 2018 Jul;22(Suppl 1):19-25. doi: 10.1007/s10461-018-2130-5. PMID 29744768